CLINICAL TRIAL: NCT00912938
Title: A Phase IV, Multi-center, Open Label, Single Arm Clinical Trial to Evaluate the Relationship of Bone Remodeling Markers for Skeletal Complications in Metastatic Breast Cancer Patients
Brief Title: Evaluate the Relationship of Bone Remodeling Markers for Skeletal Complications in Metastatic Breast Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Jae Bok Lee, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KBCSG001
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; bone remodeling markers; zoledronic acid
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zoledronic acid (Experimental): Patients with advanced breast cancer with radiographic confirmation of bone metastases. This arm will be receiving zoledronic acid administration. The primary endpoint is to find the correlation between bone turnover markers and the frequency of skeletal-related-events for one year. Skeletal related events are defined as pathologic fractures, the need for radiation therapy, orthopaedic surgery, hypercalcemia of malignancy and spinal cord compression. A total of 237 patients will be included.
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — Intravenous zoledronic acid 4mg over a minimum of 15 minutes in at least 100mls of calcium free infusion solution (0.9% sodium chloride or 5% glucose solution) every 4 weeks.
  Other Names: ZOMETA

SUMMARY:
to evaluate whether bone marker can provide the valuable predictor of skeletal complications and whether regular assessing of NTX(N-telopeptide of type I collagen) and osteocalcin can be useful in advanced breast cancer patients with bone metastasis receiving zoledronic acid.

DETAILED DESCRIPTION:
to evaluate the efficacy and safety of zoledronic acid by measuring changes in bone turnover markers

* the incidence of skeletal-related events
* time to skeletal-related events
* time to bone metastases progression
* overall survival
* the incidence of each adverse event including osteonecrosis

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced breast cancer with radiographic confirmation of bone metastases (minimum of one bone scan lesion must be confirmed as metastatic on plain radiographs or CT/MR imaging)
2. Men or women aged ≥ 18 years
3. WHO (ECOG) performance status 0-2
4. Women of child-bearing potential must be using a reliable and appropriate method of contraception
5. Urine sample taken and sent to the central laboratory for baseline Ntx analysis
6. Written informed consent.

Exclusion Criteria:

1. Bisphosphonate treatment within the 4 weeks prior to planned first study treatment
2. Abnormal renal function as evidenced by a calculated creatinine clearance < 30 ml/minute
3. Poor venous access
4. Metabolic bone disease
5. Unable to comply with study procedures, especially the reliable collection of urine samples for bone resorption marker measurements
6. Estimated life expectancy of < 6 months
7. Treatment with systemic bone seeking radioisotopes within the 3 months prior to study entry
8. Wide field (hemi-body) radiotherapy within the 3 months prior to study entry
9. Concomitant medication with drugs known to affect bone metabolism
10. Pregnancy or breast-feeding
11. Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular), or a current or prior diagnosis of osteonecrosis of the jaw (ONJ)
12. Recent (within 4 weeks of study entry*) or planned dental or jaw surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Urinary NTX and serum osteocalcin will be assessed at baseline, 3, 6, 9, and 12 months and when unexpected skeletal related events is detected. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jae Bok Lee, MD.PhD, Principal Investigator — Department of Surgery, Korea University Guro Hospital, South Korea
Locations (1):
- Department of Surgery, Korea University Guro Hospital, Seoul, South Korea